CLINICAL TRIAL: NCT01109602
Title: Yoga as a Complex Intervention for Vets With Stroke
Brief Title: Strength, Flexibility, And Balance Therapy After Stroke
Acronym: HEALTHY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRP 09-195
Record Dates: First submitted 2010-04-02; First posted 2010-04-23 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Stroke
Keywords: Stroke; accidental falls; Yoga; Blood pressure; Range of Motion; Rehabilitation; Exercise; balance; quality of life; mobility
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Pliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Yoga Group (Experimental): Yoga Group, 8 week bi-weekly in-person yoga training focused on strength, flexibility, and balance
  Yoga focused on strength, flexibility, and balance
  Interventions: Other: Yoga focused on strength, flexibility, and balance
- Arm 2: Yoga Group Plus (Experimental): Yoga Group Plus: 8 week, bi-weekly in-person yoga training focused on strength, flexibility, and balance paired with almost daily at home yoga focused on breathing and relaxation.
  Yoga focused on strength, flexibility, and balance
  Data for both yoga groups were combined for analyses as there were not any differences between these two groups.
  Interventions: Other: Yoga focused on strength, flexibility, and balance
- Arm 3: Wait list control group (No Intervention): wait-list control: will be assessed before and after 8 weeks. Will then be offered the 8 week yoga intervention.

INTERVENTIONS:
Other: Yoga focused on strength, flexibility, and balance — Participants completed 8 weeks of yoga therapy. The yoga was focused on strength, flexibility, and balance therapy after stroke to impact fear of falling, balance, mobility, QoL, and blood pressure after stroke. The in-person yoga intervention included seated, standing, and floor poses. All study participants were able to complete transfers to the floor or mat table and complete all postures and breathing exercises.
  Other Names: HEALTHY after stroke
  Arms: Arm 1: Yoga Group; Arm 2: Yoga Group Plus

SUMMARY:
Approximately 780,000 people suffer a stroke annually in the United States; 200,000 are recurrent strokes. The 17,000 veterans who suffer a stroke yearly are at great risk for a second stroke and therefore should be targeted for stroke risk factor management and prevention interventions.

Balance and fear of falling negatively impact activity and function. Decreased activity and blood pressure (BP) are important modifiable stroke risk factors. These can be addressed through a yoga exercise intervention. Yoga, like tai-chi, is old world alternative medicine that has the potential to greatly impact the lives of older adults.

DETAILED DESCRIPTION:
BACKGROUND: Approximately 780,000 people suffer a stroke annually in the United States; 200,000 are recurrent strokes. The 17,000 veterans who suffer a stroke yearly are at great risk for a second stroke and therefore should be targeted for stroke risk factor management and prevention interventions.

Balance and fear of falling negatively impact activity and function. Decreased activity and blood pressure (BP) are important modifiable stroke risk factors. These can be addressed through a yoga exercise intervention. yoga, like tai-chi, is old world alternative medicine that has the potential to greatly impact the lives of older adults.

OBJECTIVES: Our long term goal is to develop and test a yoga exercise intervention in a large VA trial for veterans who have survived a stroke. The objective of this pilot application was to obtain necessary information to support such a trial through the following specific aims: 1) determine the feasibility (including recruitment) of an 8 week yoga based intervention for veterans with stroke; 2) establish an appropriate dosing strategy for a post-stroke 8 week yoga exercise intervention for a future VA yoga implementation trial (Yoga Group, bi-weekly in-person vs Yoga Group Plus, bi-weekly in-person paired with almost daily at home yoga); and 3) estimate the effect size of yoga on variables of interest to determine the appropriate VA trial sample size.

METHODS: We completed a mixed methods study to address the feasibility, dosing strategy, and estimation of effect size for the current pilot study. We recruited 45 people with stroke to participate in the Yoga Group or Yoga Group Plus; 15 participants were wait-listed to be used as a control. A registered yoga therapist (RYT) taught all classes. Qualitative data include semi-structured interviews after completion of the intervention regarding: perceived ability to do yoga exercise; satisfaction with the yoga intervention; satisfaction with the RYT; general health benefits for the intervention; and whether they would continue yoga practice. Quantitative data included compliance and recruitment information as well as multiple standardized assessments before and after the 8 week intervention including: blood pressure readings; fear of falling; balance; balance confidence; gait and mobility assessments; and quality of life. We compared those in yoga to those wait-listed and also completed within group analyses to determine change between baseline and 8 week scores.

ELIGIBILITY:
Inclusion Criteria:

* veteran
* in the Indianapolis, IN area
* survived a stroke
* on blood pressure medication
* completed all rehabilitation
* ability to stand with or without a device
* able to speak and understand English
* a score >4 out of 6 on the short mini mental status exam (MMSE)

Exclusion Criteria:

* would not commit to the yoga intervention
* self report of: serious cardiac conditions; history of serious chronic obstructive pulmonary disease or oxygen dependence; severe weight bearing pain; a history of significant psychiatric illness; uncontrollable diabetes with recent weight loss; and current enrollment in another research trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene A. Schmid, PhD OTR MS, Principal Investigator — Richard Roudebush VA Medical Center, Indianapolis
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Schmid AA, Van Puymbroeck M, Altenburger PA, Schalk NL, Dierks TA, Miller KK, Damush TM, Bravata DM, Williams LS. Poststroke balance improves with yoga: a pilot study. Stroke. 2012 Sep;43(9):2402-7. doi: 10.1161/STROKEAHA.112.658211. Epub 2012 Jul 26. PMID 22836351

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Yoga and yoga plus groups were combined for analysis of data for Outcome Measures
Groups:
- Arm 1: Yoga Group: Yoga Group, 8 week bi-weekly in-person yoga training focused on strength, flexibility, and balance
  Yoga intervention focused on strength, flexibility, and balance therapy: Participants completed 8 weeks of yoga therapy. The yoga was focused on strength, flexibility, and balance therapy after stroke to impact fear of falling, balance, mobility, QoL, and blood pressure after stroke. The in-person yoga intervention included seated, standing, and floor poses. All study participants were able to complete transfers to the floor or mat table and complete all postures and breathing exercises.
- Arm 2: Yoga Group Plus: Yoga Group Plus: 8 week, bi-weekly in-person yoga training focused on strength, flexibility, and balance paired with almost daily at home yoga focused on breathing and relaxation. Data for both yoga groups were combined for analyses based off of data from the results.
  Yoga intervention focused on strength, flexibility, and balance therapy: Participants completed 8 weeks of yoga therapy. The yoga was focused on strength, flexibility, and balance therapy after stroke to impact fear of falling, balance, mobility, QoL, and blood pressure after stroke. The in-person yoga intervention included seated, standing, and floor poses. All study participants were able to complete transfers to the floor or mat table and complete all postures and breathing exercises.
Period: Overall Study
Arm/Group | Arm 1: Yoga Group | Arm 2: Yoga Group Plus | Arm 3: Wait List Control Group
Started | 14 | 23 | 10
Completed | 13 | 21 | 9
Not Completed | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Yoga Group | Arm 2: Yoga Group Plus | Arm 3: Wait List Control Group | Total
Number analyzed (Participants) | 14 | 23 | 10 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.33 (8.117) | 62.35 (8.526) | 60.2 (8.9) | 64.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 0 | 9
  Male | 14 | 14 | 10 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 5 | 8 | 4 | 17
  White | 8 | 14 | 6 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 23 | 10 | 47
months since stroke [Mean (Standard Deviation); unit: months] | 49.25 (44.55) | 59.13 (43.81) | 36.4 (23.6) | 51 (40.4)
type of stroke [Number; unit: participants]
  ischemic | 6 | 20 | 5 | 31
  not ischemic | 8 | 3 | 5 | 16

OUTCOME MEASURES:

1. Secondary Outcome: Balance Self-efficacy - Measured With the Activities Balance Confidence Scale
Description: The 16 item Activities-specific Balance Confidence Scale (ABC) was used to measure balance self-efficacy. The ABC is a self-report of a participant's self-efficacy in maintaining static and dynamic balance control during functional tasks. The validity and reliability of the ABC have been previously demonstrated in individuals with stroke. Scoring is 'no confidence' (0%) to 'completely confident' (100%).
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Yoga/Yoga Plus: Data for both yoga groups were combined for analyses. All participants received 8 weeks of group yoga twice a week. Participants randomized to 'yoga plus' also received an audio recording for meditation/relaxation. there were no differences between groups, thus the data were combined.
- Wait List Control Group: Participants randomized to the Wait list control group were assessed and then waited for 8 weeks for no additional intervention, just usual care. they were then assessed again 8 weeks later.
Arm/Group | Yoga/Yoga Plus | Wait List Control Group
Number analyzed (Participants) | 37 | 10
units on a scale | 66.8 (23.4) | 56.2 (25.8)

2. Primary Outcome: Balance - Measured With the Berg Balance Scale
Description: Balance was assessed with the Berg Balance Scale (BBS), a 14-item physical performance measure of static and dynamic balance found to be reliable and valid after stroke. Scoring ranges from 0-56, with higher scores indicating better balance. A score of <46 identifies an individual at risk for falls after stroke.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga/Yoga Plus | Wait List Control Group
Number analyzed (Participants) | 37 | 10
units on a scale | 46.3 (9.1) | 43.8 (6.3)

3. Secondary Outcome: Quality of Life - Measured With the Stroke Specific Quality of Life
Description: Quality of Life was measured using the validated 49 items of the Stroke Specific QoL scale (SSQoL). The SSQoL includes assessment of 12 domains: self-care; vision; language; mobility; work; upper extremity; thinking; personality; mood; family; social; and energy. Prior work indicates good psychometric properties. Higher scores indicate increased QoL. Range of scores is 13 to 65 for the total score.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga/Yoga Plus | Wait List Control Group
Number analyzed (Participants) | 37 | 10
units on a scale | 35.8 (9.1) | 33.0 (6.2)

ADVERSE EVENTS:
Time Frame: 2 month period of the intervention
Arm/Group | Arm 1: Yoga Group | Arm 2: Yoga Group Plus | Arm 3: Wait List Control Group
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/23 | 0/10
Other Adverse Events (participants affected / at risk) | 1/14 | 0/23 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Yoga Group (N=14) | Arm 2: Yoga Group Plus (N=23) | Arm 3: Wait List Control Group (N=10)
fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) — falls during the intervention time
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Yoga Group (N=14) | Arm 2: Yoga Group Plus (N=23) | Arm 3: Wait List Control Group (N=10)
hospitalization (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — aortic surgery needed, not related to intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No